CLINICAL TRIAL: NCT01658865
Title: Assessment of Esophageal Motility With Transnasal Endoscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Myung-gui Choi, prof., The Catholic University of Korea
Other Study IDs: NE-EM-001
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Esophageal Motility Disorder
MeSH Terms: conditions — Esophageal Motility Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Transnasal endoscopy: Healthy volunteers and patients with esophageal motor symptom will be enrolled and esophageal motility assessed by transnasal endoscopy according to clinical and manometric diagnosis

SUMMARY:
The purpose of this study is to assese esophageal motor function by simplified transnasal endoscopy compared with esophageal manometry.

DETAILED DESCRIPTION:
Esophageal manometry is a gold standard for diagnosis of esophageal motility disorder. However, esophageal manometry can not detect non-occulsive contraction. Endoscopic evaulation of esophageal motility is difficult becausea swallowing is nearly impossible during endoscopy. Simplified trans nasal endoscopy (E.G. ScanTM, IntroMedic Co.,Ltd.)composed with dysplay system,controller,and disposable probe with compact size.

The esophageal motor function will be assessed with both esophageal manometry and simplifed trnasnasal endoscopy in patients with esophageal motility disorder (such as achalasia) and healthy volunteer. The results of simplifed trnasnasal endoscopy is compared with the results of esophageal manometry.

ELIGIBILITY:
Inclusion Criteria:

* 1) Healthy volunteer without organic esophageal or gastric disorder 2) Patients knwon esophageal motility disorder (such as achalasia)

Exclusion Criteria:

* severe organic esophageal disorder including severe reflux esophagitis, stricture, and bleeding.
* previous opertion of esophagus or stomach
* GI bleeding, mechanical obstruction
* medication which can infulence GI motility

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with esophageal motility disorder Healthy volunteer
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-09 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Agreement of endoscopic diagnosis of esophageal motor function with manometry | one day

SECONDARY OUTCOMES:
Discomfort of simplifed transnasal endoscopy compared with esophageal manomerty estimated by the patietns | one day

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea